CLINICAL TRIAL: NCT03955250
Title: Mobile After-Care Support Intervention for Patients With Schizophrenia Following Hospitalization: Pilot RCT
Brief Title: Mobile After-Care Support App: Pilot RCT
Acronym: MACS-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1905-001; R34MH115144 (NIH)
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Results first posted 2023-08-02 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-02

CONDITIONS: Psychotic Disorder
Keywords: schizophrenia; psychosis; mHealth; psychiatric hospitalization; treatment adherence; transitions of care; coping skills; psychosocial intervention
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia; Treatment Adherence and Compliance | interventions — Amyloid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile After-Care Support (MACS) app (Experimental): All participants download the app to their mobile phone. The app runs through a third-party software platform. It is designed to provide ecological momentary assessment and intervention.
  Interventions: Behavioral: Mobile After-Care Support (MACS) app
- Mobile app attention control (Active Comparator): All participants download the app to their mobile phone. The app runs through a third-party software platform. It is designed to provide ecological momentary assessment and psychoeducation about illness.
  Interventions: Behavioral: Mobile app attention control

INTERVENTIONS:
Behavioral: Mobile After-Care Support (MACS) app — The MACS app assesses and intervenes by fostering increased treatment adherence (medication/appointments) and self-coping with illness (active, planned, problem-solving focused) to reduce symptoms and improve functioning.
  Arms: Mobile After-Care Support (MACS) app
Behavioral: Mobile app attention control — The control app provides ecological momentary assessment and psychoeducation about illness.
  Arms: Mobile app attention control

SUMMARY:
The overall aim of this program of research is to refine and test the feasibility and acceptability of a newly developed mobile device-delivered app, called Mobile After-Care Support (MACS), to improve patients' coping and treatment adherence following a hospitalization related to their psychotic-spectrum disorder. The purpose of the proposed project is to establish the feasibility, acceptability, and preliminary effects of the app. To achieve the specific aims, the investigators will conduct a pilot randomized clinical trial (n = 60), with two treatment arms: MACS vs. a mobile app attention control condition.

ELIGIBILITY:
Inclusion Criteria:

* recently hospitalized
* DSM-5 criteria for psychotic-spectrum disorder based on structured clinical interview
* 18 years or older
* prescribed antipsychotic medication upon discharge
* ability to speak and read English

Exclusion Criteria:

* substance use disorders at severe level
* planned discharge to supervised living setting or participation in formal outpatient adherence programs
* pregnancy or other medical condition contraindicating use of antipsychotic medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-05-31 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Gaudiano, PhD, Principal Investigator — Butler Hospital; Ethan Moitra, PhD, Principal Investigator — Brown University
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
Uploaded to NIMH Data Archive

REFERENCES:
- [Derived] Gaudiano BA, Ward M, Benz MB, Hughes C, Johnson JE, Moitra E. Feasibility and acceptability of a mobile intervention for patients with psychosis following psychiatric hospitalization: A pilot randomized controlled trial. Psychol Serv. 2025 May;22(2):221-231. doi: 10.1037/ser0000869. Epub 2024 Jun 6. PMID 38842850

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control
Started | 19 | 23
Completed | 17 | 16
Not Completed | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control | Total
Number analyzed (Participants) | 19 | 23 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (11.7) | 35.1 (11.1) | 34.3 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 11 | 15 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 4 | 10
  Not Hispanic or Latino | 13 | 19 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 13 | 13 | 26
  More than one race | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 23 | 42

OUTCOME MEASURES:

1. Primary Outcome: Client Satisfaction Questionnaire (CSQ)
Description: The Client Satisfaction Questionnaire is a self-report measure of patient satisfaction with treatment. The total score (sum of items) will be used and ranges from 8 to 32 with increased scores indicating greater satisfaction with treatment.
Time Frame: 1 month
Population: The number of participants analyzed is lower than the number enrolled due to missing data on this measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control
Number analyzed (Participants) | 10 | 12
score on a scale | 23.7 (4.4) | 22.5 (7.6)
Statistical Analysis 1: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Brief Psychiatric Rating Scale (BPRS)
Description: The interviewer-rated Brief Psychiatric Rating Scale is a measure of psychiatric symptom severity. The total score (sum of items) will be used to assess overall severity with scores ranging from 18 to 126 and higher scores indicating greater severity.
Time Frame: Baseline, 4 month
Population: This analysis was intent-to-treat based on all participants initially enrolled in the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control
Number analyzed (Participants) | 19 | 23
score on a scale
  Baseline | 53.1 (2.4) | 49.8 (2.2)
  4 Month | 36.4 (2.6) | 33.1 (2.6)
Statistical Analysis 1: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p < 0.05, t-test, 2 sided; time
Statistical Analysis 2: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p > 0.05, t-test, 2 sided; condition

3. Secondary Outcome: Brief Adherence Rating Scale (BARS)
Description: The Brief Adherence Rating Scale assesses the percentage of missed medication doses over the past month. The total adherence score ranges from 0% to 100% and higher scores indicate greater adherence.
Time Frame: Baseline, 4 month
Population: This analysis was intent-to-treat based on all participants initially enrolled in the study.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control
Number analyzed (Participants) | 19 | 23
units on a scale
  Baseline: number analyzed (Participants) | 19 | 20
  Baseline | 86.2 (4.8) | 83.8 (4.4)
  4 Month | 94.4 (4.9) | 92.0 (4.8)
Statistical Analysis 1: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p > 0.05, t-test, 2 sided; time
Statistical Analysis 2: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p > 0.05, t-test, 2 sided; condition

4. Secondary Outcome: Brief Cope Inventory (Brief COPE)
Description: The Brief Cope Inventory is a 28 item self-report measure of coping skills. The mean values of the 12-item dysfunctional coping subscale was used. Mean scores for the total range from 1-48 with higher scores indicating greater use of the dysfunctional coping strategies.
Time Frame: Baseline, 4 month
Population: This analysis was intent-to-treat based on all participants initially enrolled in the study.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control
Number analyzed (Participants) | 19 | 23
score on a scale
  Baseline | 28.6 (1.6) | 28.1 (1.5)
  4 Month | 24.8 (1.7) | 24.4 (1.7)
Statistical Analysis 1: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p < 0.05, t-test, 2 sided; time
Statistical Analysis 2: Comparison: Mobile After-Care Support (MACS) App vs Mobile App Attention Control; Test type: Superiority; p > 0.05, t-test, 2 sided; condition

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Mobile After-Care Support (MACS) App | Mobile App Attention Control
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/23
Serious Adverse Events (participants affected / at risk) | 11/19 | 9/23
Other Adverse Events (participants affected / at risk) | 0/19 | 0/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mobile After-Care Support (MACS) App (N=19) | Mobile App Attention Control (N=23)
Rehospitalization (Psychiatric disorders) | 9 | 9
Suicide attempt (Psychiatric disorders) | 2 | 0

LIMITATIONS AND CAVEATS:
This was a pilot RCT and therefore was designed to assess feasibility and acceptability of the intervention in preparation for a larger clinical trial. It was not powered to test comparative efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-14): https://cdn.clinicaltrials.gov/large-docs/50/NCT03955250/Prot_SAP_000.pdf